CLINICAL TRIAL: NCT04012164
Title: Viral and Microbial Circulation Between Humans, Domesticated and Wild Animals Along an Ecotone, Democratic Republic of Congo
Acronym: MICROTONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Centre National de la Recherche Scientifique, France (Other); University Paris 7 - Denis Diderot (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-085
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-08

CONDITIONS: Zoonotic Disease
Keywords: microbiome; virome; zoonotic disease; ecological gradient; human-animal relations; anthropology; social sciences
MeSH Terms: conditions — Zoonoses | interventions — Blood Specimen Collection; Contact Tracing

STUDY DESIGN:
Intervention Model Description: 2 types of participants. Human subjects participating in microbiological and anthropological study. Human subjects participating in historical and anthropological study, providing a larger context for those from whom we will collect biological samples and anthropological data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microbiological, anthropological and historical study (Experimental): 30 adult participants will be recruited to self-report daily activities and contacts with domesticated and wild animals for a five month period. Following the five months of data collection, we will collect 5ml blood and 2g stool from each participant.
  From the fifth month of investigation, an additional 30 adult participants will participate in oral anthropological, historical interviews to develop the socio-historical context of their changing activities and relations with selected domesticated and wild animals. No other intervention will be performed.
  Interventions: Biological: blood sampling; Biological: stool collection; Other: Participatory activity and contact investigation; Other: Anthropological and historical interviews

INTERVENTIONS:
Biological: blood sampling — 5ml blood sampling
Biological: stool collection — self stool collection (2g)
Other: Participatory activity and contact investigation — 30 human subjects will self-report daily activities and contacts with selected wild and domesticated animals for five months.
Other: Anthropological and historical interviews — Oral interviews on current and past practices and engagements with wild and domesticated animals will be conducted with the 30 human subjects who are recruited to self-report their activities (Participatory activity and contact investigation) and to provide blood and stool samples. Another 30 human subjects will be recruited only to participate in the same type of interviews, addressing past and present activities and relations with wild and domesticated animals.

SUMMARY:
This study will evaluate the overlap between the intestinal microbiome and virome of wild and domesticated animals and human beings living in close proximity in three sites along an ecotone (ecological gradient) in the Democratic Republic of Congo.

DETAILED DESCRIPTION:
The MICROTONE study sheds light on zoonotic disease emergence by examining social and ecological pathways facilitating microbial and viral flows between people and selected wild and domesticated animals along a gradient of ecological change in a forest-savanna mosaic in the Democratic Republic of Congo, an epicenter of zoonotic disease emergence. The investigators analyze potential viral and bacterial overlap among humans and animals and explain this overlap (or not) through social sciences and ecological analyses of human and animal mobilities, practices and contacts. This multi-disciplinary, multi-species investigation in an ecotone (a transitional ecological zone linked to zoonotic disease emergence) offers a "pre-history" of spillover and emergence, tracing an ecological zeb of virome and microbial sharing among humans and animals. It will elucidate why such microbial and viral flows occur.

To conduct this investigation,there are two human sub-studies: the social sciences participatory study; and the clinical study. The clinical study will involve 30 human subjects from whom blood and stool samples will be collected. The social sciences participatory study will involve self-collected activity and animal contact data and oral interviews among 60 human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Accept participation in study
* Residing in one of three villages selected
* In good health and able to conduct habitual daily activities
* Accept self-collection of 2g of stool
* Accept blood collection (2-2.5 ml) by a medical professional
* Accept to self-collect daily activities and contacts with selected wild and domesticated animals for five months
* Accept to participate in an anthropological-historical interview on changing practices and contacts with wild and domesticated animals

Exclusion Criteria:

* Vulnerable adults will not be included
* Women who are pregnant or nursing at the time of recruitment and inclusion will not be included.
* Adults declaring themselves ill and unable to conduct their habitual daily activities will not be included.
* Adults with a chronic illness will not be included
* Adults who have a family member already included in the study will not be included.
* Adults refusing either recording of interviews or note-taking during interviews will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Percentage of gut bacterial genera shared by included people | 2 years (March 13, 2019 to March 13, 2021)
  The investigators will evaluate the gut bacteria shared by humans on a daily basis.
Percentage of gut bacterial genera shared by selected wild animals | 2 years (March 13, 2019 to March 13, 2021)
  The investigators will evaluate the gut bacteria shared by wild animals on a daily basis.
Percentage of gut bacterial genera shared by selected domesticated animals | 2 years (March 13, 2019 to March 13, 2021)
  The investigators will evaluate the gut bacteria shared by domesticated animals living in proximity on a daily basis.
Percentage of overlap (of viral genera) between human subjects and great apes | 2 years (March 13, 2019 to March 13, 2021)
  The percentage of overlap (of viral genera) between human subjects and great apes will be measured.

SECONDARY OUTCOMES:
Description of Contact type | 2 years (March 13,2019 to March 13, 2021)
  The investigators will evaluate the type of physical contact between human beings, wild animals and domesticated animals from data collected in self-reported daily activity tool. This outcome will be measured through identified categories of physical contact. We will also estimate how contact types have changed over time through an analysis of the historical, anthropological interview data.
Contact frequency investigation | 2 years (March 13, 2019 to March 13, 2021)
  The investigators will evaluate the frequency of physical contact between human subjects and wild animals and domesticated animals from data collected in the self-reported daily activity collection tool. Frequency will be measured by the number per category of physical contact.

CONTACTS AND LOCATIONS:
Locations (1):
- INRB, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No